CLINICAL TRIAL: NCT06255249
Title: Multicenter Evaluation in Patients With MEningiomas Expressing Somatostatin Type 2 Receptors and After Failure of Standard Treatments, of the Response to Treatment With 177LUTEtium-oxodotreotide
Brief Title: Multicenter Evaluation in Patients With MEningiomas of the Response to Treatment With 177LUTEtium-oxodotreotide
Acronym: MELUTE
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Antoine VERGER, Investigator coordinator, Central Hospital, Nancy, France
Other Study IDs: 2023PI224
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Meningioma
MeSH Terms: conditions — Meningioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Meningiomas are the most common primary tumors of the central nervous system, representing more than a third of tumors.Current conventional treatments for meningioma are surgery and radiotherapy. When these treatments are no longer feasible, meningiomas are considered refractory regardless of their grade. Some meningiomas express somatostatin type 2 receptors and can be treated with lutathera. This study aims to evaluate the response to treatment in this pathology

DETAILED DESCRIPTION:
In nuclear medicine, peptide receptor radionuclide therapy with 177Lu-oxodotreotide, deploys an octreotide-like effect and appears very promising, with a preliminary progression free survival at 6 months of 94% and overall survival at 12 months of 88% in grade 1 meningiomas, and 28% with an overall survival at 12 months of 65% in grades 2 and 3 meningiomas. These results are nevertheless the result of a meta-analysis obtained from series of patients limited in number and heterogeneous in terms of type of treatment modality.

At the request of healthcare professionals and in consultation with the Advanced Accelerator Applications laboratory, the Agency of the drug security has developed a compassionate prescribing framework aimed at securing the use of Lutathera in meningiomas of all grades, expressing type 2 somatostatin in imaging of nuclear medicine, after failure of the standard treatment (surgery, radiotherapy/radio-surgery) or impossibility of carrying it out (multiple lesions, inaccessible lesions), at the suggestion of the national comitee OMEGA (April 6, 2022). This cohort has the advantage of being consistent and homogeneous in terms of type of treatment and method of administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have benefited from treatment with Lutathera® within the framework of compassionate prescription in a refractory meningioma of any grade
* Patient informed via an information and non-opposition to the use of their pseudonymized data for research purposes (research objectives clearly explained in the letters)

Exclusion Criteria:

-Patient opposition to the use of their data for this research

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients suffering from refractory meningioma of any grade who have benefited from treatment with Lutathera within the framework of compassionate prescription and who have received the information letter on the objectives of the research and who have not not opposed to the use of their data, and for which the magnetic resonance imaging will be available to be sent to a server for centralized rereading.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-10-30 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
To evaluate the response to treatment with Lutathera® in patients with meningioma expressing somatostatin type 2 receptors, and after failure of standard treatments, for whom compassionate access to this treatment has been requested. | 6 months
  Progression-free survival at 6 months (according to RANO criteria)
To evaluate the response to treatment with Lutathera® in patients with meningioma expressing somatostatin type 2 receptors, and after failure of standard treatments, for whom compassionate access to this treatment has been requested. | 12 months
  Overall survival at 12 months (according to RANO criteria)

CONTACTS AND LOCATIONS:
Overall Officials: ANTOINE VERGER, MD, PhD, Principal Investigator — CHRU Nancy
Locations (1):
- CHRU of NANCY, Vandœuvre-lès-Nancy, France